CLINICAL TRIAL: NCT01237236
Title: A phase1 Multi-center, Open Label, Dose-escalation Study of Oral LEE011 in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: A Trial of LEE011 in Patients With Advanced Solid Tumors or Lymphoma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011X2101; 2009-017017-30 (EudraCT Number)
Record Dates: First submitted 2010-11-05; First posted 2010-11-09 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2018-08

CONDITIONS: Advanced Solid Tumor; Lymphomas
Keywords: Advanced solid tumor; lymphoma
MeSH Terms: conditions — Lymphoma | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEE011 (Experimental)
  Interventions: Drug: LEE011

INTERVENTIONS:
Drug: LEE011

SUMMARY:
LEE011 is a new oral drug designed to inhibit the activity of an enzyme known as CDK4/6. CDK4/6 is involved in the process that allows both normal and cancer cells to divide and multiply. Cancer cells are often driven to divide and multiply by abnormalities that increase the activity of CDK4. Hence there is hope that blocking the activity of CDK4 may slow the growth of some cancers. LEE011 has shown anti-cancer activity in several different tumor models in animals.

Because CDK4 is important in both normal and cancerous cells, LEE011 is expected to decrease the ability of the bone marrow to make white blood cells, platelets, and red blood cells. Although these effects are expected to be reversible, they can increase the risk of infection, bleeding and fatigue.

The primary purpose of this study is to find the highest dose of LEE011 that can be safely given to adult patients with advanced solid tumors or lymphomas for which no further effective standard treatment is available. It will provide information about the side effects that may occur following treatment. The study will also possibly provide early evidence for LEE011's anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years with a histologically or cytologically confirmed diagnosis of a solid tumor or lymphoma for which no further effective standard treatment is available
2. Patients must have an ECOG performance status of 0 - 1
3. Patients enrolled in the dose expansion phase must have at least one measurable lesion as defined by RECIST criteria for solid tumors or Measurable nodal disease at baseline as defined by Cheson criteria for Lymphoma.
4. A sufficient interval must have elapsed between the last dose of prior anti-cancer therapy (including cytotoxic and biological therapies and major surgery) and enrollment in this study, to allow the effects of prior therapy to have abated:

   * Cytotoxic chemotherapy: ≥ the duration of the cycle of the most recent treatment regimen (a minimum of 2 weeks for all regimens, except 6 weeks for nitrosoureas and mitomycin-C).
   * Biologic therapy (e.g., antibodies): ≥ 4 weeks.
5. Patients must have adequate organ function, as defined by the following parameters:

   * Bone marrow: Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L, Hemoglobin (Hgb) ≥ 9 g/dL, Platelets ≥ 100 x 109/L
   * Hepatic function: Serum total bilirubin ≤ 1.5 x ULN (upper limit of normal); AST (SGOT) and ALT (SGPT) ≤ 3 x ULN, except in patients with tumor involvement of the liver who must have AST and ALT ≤ 5 x ULN
   * Renal function: Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 40 ml/min, Serum potassium, magnesium and calcium must be within normal limits

Exclusion Criteria:

1. Patients with primary central nervous system tumors or brain metastases. However, if radiation therapy and/or surgery has been completed and serial evaluation by CT (with contrast enhancement) or MRI over a minimum of 3 months demonstrates the disease to be stable and if the patient remains asymptomatic, then the patient may be enrolled. Such patients must have no need for treatment with steroids or anti-epileptic medications.
2. Impairment of gastro-intestinal (GI) function or GI disease that may significantly alter the absorption of LEE011 such as patients with a history of GI surgery which may result in intestinal blind loops and patients with clinically significant gastroparesis, unresolved nausea, vomiting, or diarrhea of CTCAE grade > 1
3. Prior hematopoietic stem cell or bone marrow transplantation
4. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   * LVEF <45% as determined by MUGA or echo
   * Complete left bundle branch block
   * Obligate use of a cardiac pacemaker or implantable cardioverter defibrillator
   * Congenital long QT syndrome or family history of unexpected sudden cardiac death
   * History or presence of ventricular tachyarrhythmia
   * Presence of unstable atrial fibrillation (ventricular response > 100 bpm
   * Clinically significant resting bradycardia
   * QTcF >450 ms for males and >470 ms for females on screening ECG
   * Right bundle branch block and left anterior hemiblock (bifascicular block)
   * Angina pectoris ≤ 3 months prior to dosing with study drug
   * Acute MI ≤ 3 months prior to dosing with study drug
   * Other clinically significant heart disease
5. Acute myocardial infarction or angina pectoris ≤ 3 months prior to starting study drug
6. Patients with concurrent severe and/or uncontrolled concurrent medical conditions that could compromise participation in the study (e.g. uncontrolled hypertension and/or diabetes mellitus, clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection).

Known diagnosis of HIV or hepatitis C

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2010-12-21 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures: Maximum tolerated dose of LEE011 when administered orally once daily, as assessed by Frequency of DLTs as a function of LEE011 dose | 12 month

SECONDARY OUTCOMES:
Safety and tolerability of LEE011, as assessed by grade and frequency of Adverse events, serious adverse events, and changes in lab values, vital signs and ECGs. | 18 months
The pharmacokinetics (PK) of LEE011 (AUC inf, Cmax, Tmax, T1/2) | 18 months
Any pharmacodynamic activity of LEE011 treatment, as assessed by changes from baseline in biomarkers associated with the pharmacologic activity of LEE011 | 18 months
Antitumor activity that may be associated with LEE011 treatment, as assessed by CT/MRI Response Evaluation Criteria for Solid Tumors (RECIST) Criteria v1.0 or Cheson Criteria 2007 for lymphomas. | 18 months
Relationship between QTc prolongation and exposure to LEE011 and/or any of its relevant metabolites. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (4):
  - Dana Farber Cancer Institute DFCI, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center SC, Ann Arbor, Michigan
  - Memorial Sloan Kettering MSKCC (2), New York, New York
  - Sarah Cannon Research Institute DeptofSarahCannonRes.Inst. (2), Nashville, Tennessee
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Utrecht, Netherlands

REFERENCES:
- [Derived] Ji Y, Yartsev V, Quinlan M, Serra P, Wang Y, Chakraborty A, Miller M. Justifying Ribociclib Dose in Patients with Advanced Breast Cancer with Renal Impairment Based on PK, Safety, and Efficacy Data: An Innovative Approach Integrating Data from a Dedicated Renal Impairment Study and Oncology Clinical Trials. Clin Pharmacokinet. 2023 Mar;62(3):493-504. doi: 10.1007/s40262-022-01206-2. Epub 2023 Feb 17. PMID 36800111
- See also: Results for CLEE011X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17048